CLINICAL TRIAL: NCT01950390
Title: A Randomized Phase II Trial of Ipilimumab With or Without Bevacizumab in Patients With Unresectable Stage III or Stage IV Melanoma
Brief Title: Ipilimumab With or Without Bevacizumab in Treating Patients With Stage III-IV Melanoma That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-01732; NCI-2013-01732 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E3612; ECOG-E3612; E3612 (Other: ECOG-ACRIN Cancer Research Group); E3612 (Other: CTEP); U10CA021115 (NIH); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Results first posted 2024-04-25 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Stage IIIC Cutaneous Melanoma AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7; Unresectable Melanoma
MeSH Terms: conditions — Melanoma | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Ipilimumab; CTLA-4 Antigen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (ipilimumab) (Active Comparator): INDUCTION THERAPY: Patients receive ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Beginning cycle 8, patients receive ipilimumab IV over 90 minutes on day 1. Cycles repeat every 12 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab
- Arm B (ipilimumab and bevacizumab) (Experimental): INDUCTION THERAPY: Patients receive ipilimumab IV over 90 minutes and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive bevacizumab as in Induction Therapy. Beginning cycle 8, patients also receive ipilimumab IV over 90 minutes on day 1. Cycles repeat every 12 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Biological: Ipilimumab

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
  Arms: Arm B (ipilimumab and bevacizumab)
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy

SUMMARY:
This randomized phase II trial studies how well ipilimumab with or without bevacizumab works in treating patients with stage III-IV melanoma that cannot be removed by surgery. Immunotherapy with monoclonal antibodies, such as ipilimumab and bevacizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare overall survival for patients receiving ipilimumab plus bevacizumab versus ipilimumab alone.

SECONDARY OBJECTIVES:

I. To evaluate the progression free survival, response rate and safety in patients receiving ipilimumab plus bevacizumab versus ipilimumab alone.

II. To evaluate the utility of immune related response criteria (irRC) in patients receiving ipilimumab plus bevacizumab versus ipilimumab alone.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A:

INDUCTION THERAPY: Patients receive ipilimumab intravenously (IV) over 90 minutes on day 1. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Beginning cycle 8, patients receive ipilimumab IV over 90 minutes on day 1. Cycles repeat every 12 weeks in the absence of disease progression or unacceptable toxicity.

ARM B:

INDUCTION THERAPY: Patients receive ipilimumab IV over 90 minutes and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients receive bevacizumab as in Induction Therapy. Beginning cycle 8, patients also receive ipilimumab IV over 90 minutes on day 1. Cycles repeat every 12 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status: 0 or 1
* Untreated or previously received one treatment regimen for measurable unresectable stage III or stage IV melanoma (American Joint Committee on Cancer [AJCC] 2010) (for BRAF wild-type, and regardless of human leukocyte antigen [HLA] type); untreated or previously received up to two treatment regimens for measurable unresectable stage III or stage IV melanoma (AJCC 2010) (for BRAF mutant, and regardless of HLA type; if 2 prior regimens, one should be a BRAF inhibitor); this does not include any therapies given in the adjuvant setting
* Prior treatment (chemotherapy [chemo], radiation, hormone, and immune therapies) must be completed > 4 weeks prior to randomization (> 6 weeks prior to randomization for nitrosoureas, mitomycin C, and checkpoint inhibitors)
* Patients who received prior therapy with anthracyclines should have a baseline multigated acquisition scan (MUGA) or echocardiogram (echo) with a normal ejection fraction within 28 days prior to randomization
* Patients must have recovered from any acute toxicity associated with prior therapy by the start of study treatment
* Women must not be pregnant or breast-feeding due to the unknown effects on the fetus or infant; all females of childbearing potential must have a blood test or urine study within 2 weeks prior to randomization to rule out pregnancy; a female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* All sites of disease must be evaluated within 4 weeks prior to randomization; patients must have measurable disease
* White blood cell (WBC) >= 2000/uL (obtained within 4 weeks prior to randomization)
* Absolute neutrophil count (ANC) >= 1000/uL (obtained within 4 weeks prior to randomization)
* Platelets >= 75 x 10^3/uL (obtained within 4 weeks prior to randomization)
* Hemoglobin >= 9 g/dL (obtained within 4 weeks prior to randomization)
* Creatinine =< 2.0 x upper limit of normal (ULN) (obtained within 4 weeks prior to randomization)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x ULN for patients without liver metastases and =< 5 x ULN for patients with liver metastases (obtained within 4 weeks prior to randomization)
* Serum bilirubin =< 2.0 x ULN (except patients with Gilbert's syndrome, who must have a total bilirubin less than 3.0 mg/dL) (obtained within 4 weeks prior to randomization)
* Patients BRAF mutation status must be known
* No concomitant therapy with any of the following: interleukin (IL) 2, interferon, or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigational therapies; or chronic use of systemic corticosteroids; must have been discontinued >= 4 weeks prior to randomization
* No infection with human immunodeficiency virus (HIV); due to the mechanism of action of ipilimumab and bevacizumab, activity and side effects in an immune compromised patient are unknown
* No active infection with hepatitis B
* No active or chronic infection with hepatitis C
* Patients are ineligible if they have any history of central nervous system (CNS) metastases
* Patients are ineligible if they have a history of any other malignancy from which the patient has been disease-free for less than 2 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix
* Patients are ineligible if they have a history of autoimmune disease, as follows: patients with a history of inflammatory bowel disease are excluded from this study as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's granulomatosis]); patients with motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre syndrome and myasthenia gravis) are excluded; patients with a history of autoimmune thyroiditis are eligible if their current thyroid disorder is treated and stable with replacement or other medical therapy
* Patients are ineligible if they have an active infection
* Patients are ineligible if they have a history of prior treatment with ipilimumab, bevacizumab, or prior tumor CD137 agonist or CTLA-4 inhibitor or agonist; patients may be treatment naive or have had one prior systemic therapy for metastatic disease as outlined in the eligibility criteria; patients may have received PD-1 or PD-L1 as per current protocol eligibility, although they are not currently commercially approved in the front line setting
* Patients are ineligible if they have a history of any underlying medical or psychiatric conditions or require any medications or treatment that in the opinion of the principal investigator may interfere with compliance, make the administration of study drug hazardous or obscure the interpretation of adverse events, such as a condition associated with frequent diarrhea
* Patients are ineligible if they have any concurrent medical condition requiring the use of systemic steroids; (use of inhaled or topical steroids is acceptable)
* Patients are ineligible if they have inadequately controlled hypertension (defined as systolic blood pressure > 150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
* Patients are excluded if they have any prior history of hypertensive crisis or hypertensive encephalopathy
* Patients are excluded if they have New York Heart Association (NYHA) grade II or greater congestive heart failure
* Patients are excluded if they have a history of myocardial infarction or unstable angina within 6 months prior to randomization
* Patients are excluded if they have a history of stroke or transient ischemic attack within 6 months prior to randomization
* Patients are excluded if they have known significant vascular disease (e.g., aortic aneurysm, aortic dissection)
* Patients are excluded if they have symptomatic peripheral vascular disease
* Patients are excluded if they have evidence of bleeding diathesis or coagulopathy
* Patients are excluded if they have had a surgical procedure or a significant traumatic injury within 28 days prior to randomization
* Patients are excluded if they have had a biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to randomization
* Patients are excluded if they have history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to randomization
* Patients are excluded if they have a non-healing wound or ulcer
* Patients are excluded if they have proteinuria at screening as demonstrated by either:

  * Urine dipstick for proteinuria >= 2+ (patients discovered to have >= 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate =< 1 g of protein in 24 hours to be eligible) OR
  * Urine protein: creatinine (UPC) ratio >= 1.0 at screening; for UPC ratio > 1, a 24 hour urine protein should be obtained and the level should be < 1000 mg; NOTE: urine protein should be screened by urine analysis for UPC ratio; a UPC ratio of 1 is roughly equivalent to a 24-hour urine protein of 1 g
* Patients must not have known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Patients are excluded if they have a history of hemoptysis (bright red blood of 1/2 teaspoon or more per episode) within 3 months prior to randomization
* Patients are excluded if they have current, ongoing treatment with full-dose warfarin or its equivalent (i.e., unfractionated and/or low molecular weight heparin); subjects should have not taken full-dose warfarin or equivalent for at least 2 weeks prior to randomization
* Patients are excluded if they have current or recent (within 10 days of enrollment) use of aspirin (> 325 mg/day) or chronic use of other non-steroidal anti-inflammatory drugs (NSAIDs)
* Patients are excluded if they use medications that inhibit platelet function (e.g., dipyridamole, epoprostenol, eptifibatide, clopidogrel, cilostazol, abciximab, ticlopidine, and ibuprofen and related compounds) unless subject has been off treatment for at least 2 weeks prior to randomization
* Patients are excluded if they have known involvement of melanoma within the gastrointestinal tract
* Patients are excluded for any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 1 month before or after any dose of ipilimumab)
* Women of childbearing potential and sexually active males must agree to practice abstinence or use an accepted and effective method of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2014-01-24 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2025-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank S Hodi, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (482):
- United States (482):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - UChicago Medicine Comprehensive Cancer Center - Saint Joseph Hospital, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - UChicago Medicine AdventHealth Cancer Institute Hinsdale, Hinsdale, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - JCHC McCreery Cancer Center, Fairfield, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Covington, Covington, Louisiana
  - Mary Bird Perkins Cancer Center - Houma, Houma, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Faith Regional Health Services Carson Cancer Center, Norfolk, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Urology Cancer Center PC, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Dartmouth Cancer Center - Manchester, Manchester, New Hampshire
  - Dartmouth Cancer Center - Nashua, Nashua, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Hematology Oncology Associates of CNY at Camillus, Camillus, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Salem Hospital, Salem, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Lakeview Medical Center-Marshfield Clinic, Rice Lake, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on December 13, 2013, and closed to accrual on September 25, 2017, with a final accrual of 169 patients.
Groups:
- Arm A (Ipilimumab): INDUCTION THERAPY: Patients receive ipilimumab 3mg/kg IV over 90 minutes on day 1. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Beginning cycle 8, patients receive ipilimumab 3mg/kg IV over 90 minutes on day 1 of every 4 cycles (12 weeks) in the absence of disease progression or unacceptable toxicity.
  Ipilimumab: Given IV
- Arm B (Ipilimumab and Bevacizumab): INDUCTION THERAPY: Patients receive ipilimumab 3mg/kg IV over 90 minutes and bevacizumab 15mg/kg IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive bevacizumab as in Induction Therapy. Beginning cycle 8, patients also receive ipilimumab 3mg/kg IV over 90 minutes on day 1 of every 4 cycles (12 weeks) in the absence of disease progression or unacceptable toxicity.
  Bevacizumab: Given IV
  Ipilimumab: Given IV
Period: Overall Study
Arm/Group | Arm A (Ipilimumab) | Arm B (Ipilimumab and Bevacizumab)
Started | 85 | 84
Started Treatment | 82 | 82
Completed | 1 | 0
Not Completed | 84 | 84
Not completed — Never started treatment | 3 | 2
Not completed — Disease progression | 45 | 52
Not completed — Adverse Event | 22 | 16
Not completed — Death | 5 | 3
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Alternative therapy | 0 | 3
Not completed — Complicating disease | 1 | 0
Not completed — On treatment | 1 | 0
Not completed — Symptomatic deterioration | 2 | 1
Not completed — Physician Decision | 0 | 4
Not completed — Lack of clinical benefit | 0 | 1
Not completed — Maintained PR and moved to observation only | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Ipilimumab) | Arm B (Ipilimumab and Bevacizumab) | Total
Number analyzed (Participants) | 85 | 84 | 169
Age, Continuous [Median (Full Range); unit: years] | 65 [26 to 91] | 65 [36 to 87] | 65 [26 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 43 | 71
  Male | 57 | 41 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 80 | 79 | 159
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 81 | 80 | 161
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS distributions will be estimated using the Kaplan-Meier method. The distribution of OS will be compared using the stratified log rank test with one-sided overall type I error rate of 0.100 (adjusting for the one interim analysis) and the hazard ratio of OS will be estimated using the stratified Cox proportional hazard model and one-sided 90% repeated confidence interval will be constructed.
Time Frame: Time from randomization to death from any cause, assessed up to 5 years
Population: All enrolled patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Ipilimumab) | Arm B (Ipilimumab and Bevacizumab)
Number analyzed (Participants) | 85 | 84
months | 20.4 [13.2 to 31.6] | 20.1 [13.3 to 27.6]
Statistical Analysis 1: Comparison: Arm A (Ipilimumab) vs Arm B (Ipilimumab and Bevacizumab); Test type: Superiority; p = 0.383, Log Rank — One-sided; Stratification factors of BRAF mutation status (wild type/mutation) and prior therapy (yes/no) were used in the stratified analysis; Hazard Ratio (HR) = 0.94, 90% CI 1-sided [upper limit 1.23] — One-sided 90% Repeated Confidence Interval for Hazard Ratio with Arm A as Reference

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Evaluated based on international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Progression is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: The appearance of one or more new lesions is also considered progression). Will be estimated using the Kaplan-Meier method. PFS distributions will be compared using the log-rank test.
Time Frame: Time from randomization to disease progression or death (whichever occurs first), assessed up to 5 years
Population: All enrolled patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Ipilimumab) | Arm B (Ipilimumab and Bevacizumab)
Number analyzed (Participants) | 85 | 84
months | 2.8 [2.6 to 3.1] | 4.4 [2.9 to 6.2]
Statistical Analysis 1: Comparison: Arm A (Ipilimumab) vs Arm B (Ipilimumab and Bevacizumab); Test type: Superiority; p = 0.358, Log Rank — Two-sided; Stratified Log rank test; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.61 to 1.20]

3. Secondary Outcome: Clinical Response Rate
Description: Clinical Response Rate is defined as the percentage of patients whose tumors have a complete response (CR) or partial response (PR) to treatment. Defined by Response Evaluation Criteria in Solid Tumors version 1.1. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 5 years
Population: All enrolled patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Ipilimumab) | Arm B (Ipilimumab and Bevacizumab)
Number analyzed (Participants) | 85 | 84
percentage of participants | 11.8 [4.9 to 18.6] | 15.5 [7.7 to 23.2]
Statistical Analysis 1: Comparison: Arm A (Ipilimumab) vs Arm B (Ipilimumab and Bevacizumab); Test type: Superiority; p = 0.482, Chi-squared — Two-sided

4. Secondary Outcome: Incidence of Adverse Events (AE)
Description: Treatment-related grade 3-5 worst degree AEs rate. Defined using the Common Terminology Criteria for Adverse Events version 4.0 criteria (version 5.0 effective April 1,2018).
Time Frame: Up to 90 days after completion of study treatment, up to 5 years post-registration.
Population: All patients who received treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Ipilimumab) | Arm B (Ipilimumab and Bevacizumab)
Number analyzed (Participants) | 82 | 82
percentage of participants | 39 [28.4 to 49.6] | 58 [47.3 to 68.7]

5. Secondary Outcome: Immune-related (ir) Responses Rate (Ir-CR+Ir-PR)
Description: Assessed using the utility of irRC. Immune-Related Complete Response (irCR): Complete disappearance of all tumor lesions (target and non-target together with no new measurable/unmeasurable lesions) for at least 4 weeks from the date of documentation of complete response. Immune-Related Partial Response (irPR): The sum of the products of the two largest perpendicular diameters of all target lesions is measured and captured as the SPD baseline. At each subsequent tumor assessment, the SPD of the two largest perpendicular diameters of all target lesions and of new measurable lesions are added together to provide the Immune Response Sum of Product Diameters (irSPD). A decrease, relative to baseline of the irSPD compared to the previous SPD baseline, of 50% or greater is considered an immune Partial Response (irPR).
Time Frame: Up to 5 years
Population: Patients with reported IR responses
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Ipilimumab) | Arm B (Ipilimumab and Bevacizumab)
Number analyzed (Participants) | 39 | 52
percentage of participants | 17.9 [7.5 to 33.5] | 17.3 [8.2 to 30.3]
Statistical Analysis 1: Comparison: Arm A (Ipilimumab) vs Arm B (Ipilimumab and Bevacizumab); Test type: Superiority; p = 0.937, Chi-squared — Two-sided

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment, up to 5 years.
Description: All 169 enrolled in the trial were monitored for mortality. Only patients who started protocol therapy reported adverse events data. Serious adverse events are defined as grade 3 or higher treatment-related adverse events.
Arm/Group | Arm A (Ipilimumab) | Arm B (Ipilimumab and Bevacizumab)
All-Cause Mortality (participants affected / at risk) | 57/85 | 54/84
Serious Adverse Events (participants affected / at risk) | 32/82 | 48/82
Other Adverse Events (participants affected / at risk) | 72/82 | 77/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Ipilimumab) (N=82) | Arm B (Ipilimumab and Bevacizumab) (N=82)
Anemia (Blood and lymphatic system disorders) | 1 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 4 | 8
Gait disturbance (General disorders) | 0 | 1
Sudden death NOS (General disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 5
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 3 | 2
Hypothyroidism (Endocrine disorders) | 0 | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Colitis (Gastrointestinal disorders) | 5 | 5
Colonic perforation (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 14 | 6
Mucositis oral (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Rectal fistula (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Autoimmune disorder (Immune system disorders) | 3 | 0
Lung infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 5 | 2
Aspartate aminotransferase increased (Investigations) | 3 | 2
Blood bilirubin increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 4 | 3
Lymphocyte count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Serum amylase increased (Investigations) | 1 | 1
Investigations - Other, specify (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 6
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 4 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 2
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Hematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 29
Hypotension (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Ipilimumab) (N=82) | Arm B (Ipilimumab and Bevacizumab) (N=82)
Anemia (Blood and lymphatic system disorders) | 10 | 13
Chills (General disorders) | 7 | 7
Edema limbs (General disorders) | 2 | 10
Fatigue (General disorders) | 46 | 50
Fever (General disorders) | 7 | 8
Pain (General disorders) | 1 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 34 | 27
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 35 | 30
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 5 | 5
Adrenal insufficiency (Endocrine disorders) | 2 | 5
Hypothyroidism (Endocrine disorders) | 7 | 15
Endocrine disorders - Other, specify (Endocrine disorders) | 1 | 6
Abdominal pain (Gastrointestinal disorders) | 13 | 12
Constipation (Gastrointestinal disorders) | 4 | 7
Diarrhea (Gastrointestinal disorders) | 28 | 33
Mucositis oral (Gastrointestinal disorders) | 4 | 7
Nausea (Gastrointestinal disorders) | 16 | 19
Vomiting (Gastrointestinal disorders) | 6 | 9
Alanine aminotransferase increased (Investigations) | 17 | 21
Alkaline phosphatase increased (Investigations) | 6 | 6
Aspartate aminotransferase increased (Investigations) | 23 | 20
Creatinine increased (Investigations) | 5 | 10
Lipase increased (Investigations) | 10 | 14
Platelet count decreased (Investigations) | 4 | 8
Serum amylase increased (Investigations) | 6 | 8
Weight loss (Investigations) | 7 | 12
Investigations - Other, specify (Investigations) | 4 | 13
Anorexia (Metabolism and nutrition disorders) | 15 | 23
Dehydration (Metabolism and nutrition disorders) | 6 | 8
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 9
Hyperuricemia (Metabolism and nutrition disorders) | 2 | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 7
Hypokalemia (Metabolism and nutrition disorders) | 6 | 5
Hyponatremia (Metabolism and nutrition disorders) | 7 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 9
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 8 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 6
Dizziness (Nervous system disorders) | 4 | 9
Headache (Nervous system disorders) | 9 | 21
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Chronic kidney disease (Renal and urinary disorders) | 0 | 5
Proteinuria (Renal and urinary disorders) | 4 | 25
Hypertension (Vascular disorders) | 10 | 39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/90/NCT01950390/Prot_SAP_000.pdf